CLINICAL TRIAL: NCT01470625
Title: Improving Quality of Care for the Dying Patient in Hospice: A Quasi Experimental Trial in Liguria Region
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regional Palliative Care Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: LCP-I LIG
Record Dates: First submitted 2011-10-21; First posted 2011-11-11 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: End-of-Life
Keywords: Dying; Patients; Hospice; Liverpool Care Pathways
MeSH Terms: conditions — Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LCP Program (Other): The LCP Program is continuous quality improvement program of end-of-life care implemented in hospice
  Interventions: Other: LCP Program

INTERVENTIONS:
Other: LCP Program — The LCP Program is continuous quality improvement program of end-of-life care implemented in hospice

SUMMARY:
This is a before-after phase II study, according to the Medical Research Council framework, investigating the feasibility of introducing the Liverpool Care Pathway for the dying patient (LCP) in 5 Ligurian hospices.

ELIGIBILITY:
Inclusion Criteria:

* All patients deceased in the hospice during the evaluation period
* Approval of ethics committee

Exclusion Criteria:

* Prior use of LCP in the hospice
* Deceased was a relative of a hospice member of staff

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2010-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
feasibility of LCP implementation | 6 months after the end of LCP implementation
  measured as proportion of hospices that complete the experimental phase of introducing the LCP Program and maintain the program in the 6 months subsequent the process of experimental LCP implementation

SECONDARY OUTCOMES:
quality of information provided to patients and to family | 2-4 months after the patient's death
  measured with the scale 1 (Informing and promoting shared decision making) from the Toolkit After-death bereaved family member interview (Teno 2001). The Toolkit will be administered to non-professional caregivers 2-4 months after the patient's death
Level of advanced care planning among patients | 2 - 4 months after the patient's death
  measured with the scale 2 (Encouraging advance care planning) from the Toolkit After-death bereaved family member interview (Teno 2001). The Toolkit will be administered to non-professional caregivers 2-4 months after the patient's death
Provision of care focusing on patient's individual needs. | 2 - 4 months after the patient's death
  measured with the scale 3 (Focus on individual) from the Toolkit After-death bereaved family member interview (Teno 2001). The Toolkit will be administered to non-professional caregivers 2-4 months after the patient's death
Quality of emotional support to family members before an after the patient's death | 2 - 4 months after the patient's death
  measured with the scale 4 (Attending to the emotional and spiritual needs of the family) from the Toolkit After-death bereaved family member interview (Teno 2001). The Toolkit will be administered to non-professional caregivers 2-4 months after the patient's death
Level of care coordination | 2 - 4 months after the patient's death
  measured with the scale 5 (Providing coordination of care) from the Toolkit After-death bereaved family member interview (Teno 2001). The Toolkit will be administered to non-professional caregivers 2-4 months after the patient's death
Family support levels | 2 - 4 months after the death of the patient
  measured with the scale 6 (Supporting the self-efficacy of the family) from the Toolkit After-death bereaved family member interview (Teno 2001). The Toolkit will be administered to non-professional caregivers 2-4 months after the patient's death
Appropriateness of therapeutic and diagnostic procedures | the last 3 days of life
  measured with a specific tool in which all diagnostic and therapeutic procedures and drugs administered to the patient during the last 3 days of life are reported
Overall quality of care experience for patients and family | 2 - 4 months after the death of the patient
  measured with the scale 7 (Overall quality of care provided to patients and family) from the Toolkit After-death bereaved family member interview (Teno 2001). The Toolkit will be administered to non-professional caregivers 2-4 months after the patient's death
Quality of communication between General Practitioner and hospice | an expected average of 2 months after the patient's death
  measured with a telephonic interview

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Costantini, Study Chair — IRCCS AOU San Martino- IST
Locations (5):
- Italy (5):
  - Hospice ASL 4, Chiavari, Genova
  - Hospice Gigi Ghirotti "Albaro", Genova
  - Hospice Gigi Ghirotti "Bolzaneto", Genova
  - Hospice ASL1 Liguria, Imperia
  - CENTRO MISERICORDIA" SANTA M.G.ROSSELLO. Ist.Figlie Ns Signora Misericordia, Savona